CLINICAL TRIAL: NCT02566980
Title: The Role of Kynurenine Pathway Metabolites in Perinatal Depression and Suicidality
Brief Title: Biological Triggers of Depression in Pregnancy
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Collaborators: Pine Rest Christian Mental Health Services (Other); Van Andel Research Institute (Other); Corewell Health West (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lena Brundin, Associate Professor, Division of Psychiatry and Behavioral Medicine, Michigan State University
Other Study IDs: 14-458M; 1R01MH104622-01 (NIH)
Record Dates: First submitted 2015-09-25; First posted 2015-10-02 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Depression and Suicide; Mood Disorders; Other Perinatal Conditions
Keywords: depression; mood disorder; post-partum depression; suicidality; post-partum suicidality; perinatal depression; perinatal mood disorder; inflammation; kynurenine pathway; glutamate
MeSH Terms: conditions — Depression; Suicide; Mood Disorders; Depression, Postpartum; Suicidal Ideation; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adult Blood Cord Blood Placenta
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pre-partum: 130 pregnant women will be enrolled in first trimester. Healthy women or those with any degree of depressive symptoms are eligible. Blood samples and psychiatric assessments will take place once every trimester and once in the post-partum. At delivery placenta will be collected. Enrollment takes place at Spectrum Health Ob/gyn out-patient clinics in Grand Rapids, Michigan.
- Post-partum: 50-100 women experiencing perinatal depression with and without suicidality will be enrolled from a partial hospitalization program, the Mother and Baby unit as well as outpatient clinics at Pine Rest Christian Mental Health Services, Grand Rapids, Michigan.

SUMMARY:
The goal of the study is to define and measure biological processes that contribute to the underlying pathophysiologic process of peri-partum depression to be used for identifying those at risk for developing it. This knowledge may also generate novel drug targets for peripartum depression that may be applicable to other types of depression.

DETAILED DESCRIPTION:
This study analyses the role of inflammation and metabolites of inflammation in perinatal depression. Psychiatric assessments of depression and suicidality will be compared to blood levels of two metabolites of inflammation, quinolinic acid (QUIN) and picolinic acid (PIC), that might regulate nerve cell communication. The levels of these metabolites are regulated by kynurenine pathway enzymes.

Psychiatric symptoms, inflammatory cytokines and levels of the metabolites will be measured throughout pregnancy. Additionally, the investigators are gathering placentas at delivery and determining the degree of inflammation in the tissue in the investigators' laboratory. Inflammatory biomarkers, antibody titers, and key kynurenine pathway enzymes and metabolites from pre- and post partum women, placenta, and cord blood will be measured.

ELIGIBILITY:
Inclusion Criteria

Pre-partum cohort:

* All races and national origins of pregnant females.
* Age 18 and older.
* English speaking.
* Able to give informed consent.
* Able to comply with study procedures.

Exclusion Criteria

Pre-partum cohort:

* Non-pregnant females
* Patients with psychotic symptoms and/or severe cognitive impairment that interfere with their ability to give informed consent or to complete study assessments.
* Patients that cannot read and write in English as research measures used have only been validated in English speaking populations.
* Patients that have blood-borne chronic infections including hepatitis B, C, or HIV as established at routine pregnancy blood screens; they will be excluded as the laboratory facilities do not approve processing of their tissue for safety reasons.
* Patients who have any schizophrenia spectrum disorder or bipolar disorder type 1 (based on self report and SCID interview); these patients will be excluded as the neurobiology of these disorders are different from peripartum depression.
* Patients who report ongoing substance abuse or dependence (in the past 3 months).

Inclusion criteria

Post-partum cohort:

* All races and national origins of females who delivered a child vaginally or by caesarian section up to 6 months prior to enrollment.
* Age 18 and older.
* Edinburgh Perinatal Depression Rating Scale score of 10 and above and/or endorsed suicide ideation on the CSSRS.
* Depressive symptoms which began or worsened (if already present) during pregnancy or up to 4 weeks post-partum.
* Able to give informed consent.
* Able to comply with and complete study procedures.
* English speaking.

Exclusion criteria

Post-partum cohort:

* Patients with psychotic symptoms and/or severe cognitive impairment that interfere with their ability to give informed consent or to complete study assessments.
* Patients who cannot read and write in English as research measures used have only been validated in English speaking populations.
* Patients that have blood-borne chronic infections including hepatitis B, C, or HIV; as established at their routine pregnancy blood screens.
* Patients who have any schizophrenia spectrum disorder or bipolar type 1 (based on the self report and SCID interview).
* Patients who report ongoing substance abuse or dependence (past 3 months).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant females age 18 and older, psychiatrically healthy or depressed; post-partum females experiencing perinatal depression with and without suicide ideation.
Sampling Method: Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Change in activity of the enzyme aminocarboxymuconate semialdehyde decarboxylase ACMSD in blood during pregnancy | Up to pregnancy week 13 (1st sample), up to week 25 (second sample) and up to delivery (3rd sample) and post-partum (4th sample, within 6 months after delivery)
  Blood levels of quinolinic acid and picolinic acid (product of ACMSD) at three timepoints during pregnancy and one time-point after pregnancy
Activity of the enzyme aminocarboxymuconate semialdehyde decarboxylase ACMSD in placenta | At delivery
  Placenta levels of quinolinic acid and picolinic acid
Increase in depressive symptoms | Up to pregnancy week 13 (1st assessment), up to week 25 (second assessment) and up to delivery (3rd assessment) and post-partum (4th assessment, within 6 months after delivery)
  Assessment of depressive symptoms by means of the Edinburgh Postnatal Depression Scale
Suicidal symptoms | Post-partum (within 6 months after delivery).
  Assessment of suicidal symptoms by means of the Columbia Suicide Severity Rating Scale

SECONDARY OUTCOMES:
Change in blood inflammation | Up to pregnancy week 13 (1st sample), up to week 25 (second sample) and up to delivery (3rd sample) and post-partum (4th sample, within 6 months after delivery)
  Analysis of the inflammatory cytokine IL-6 in blood
Placenta inflammation | At delivery
  Analysis of the expression of the inflammatory cytokine IL-6 in placental tissue

CONTACTS AND LOCATIONS:
Overall Officials: Lena Brundin, MD, PhD, Principal Investigator — Michigan State University, Van Andel Research Institute
Locations (3):
- United States (3):
  - Spectrum Health System, Grand Rapids, Michigan
  - Van Andel Research Institute, Grand Rapids, Michigan
  - Pine Rest Christian Mental Health Services, Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Institute of Mental Health (NIMH), Statistics Use of Mental Health Services and Treatment among Adults. Availabe on-line at http://www.nimh.nih.gov/statistics/3USE_MT_ADULT.shtml.
- [Background] World Health Organization (WHO). What Is Depression. Available on-line at http://www.who.int/mental_health/management/depression/definition/en/
- [Background] First MB, Spitzer RL, Gibbon M, Williams JBW. Structured Clinical Interview for DSM-IV Axis I Disorders - Patient Edition (SCID-I/P, Version 2.0), Biometrics Research Department, New York State Psychiatric Institute, 1995.
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of self-reported postpartum depressive symptoms--17 states, 2004-2005. MMWR Morb Mortal Wkly Rep. 2008 Apr 11;57(14):361-6. PMID 18401329
- [Background] Dietz PM, Williams SB, Callaghan WM, Bachman DJ, Whitlock EP, Hornbrook MC. Clinically identified maternal depression before, during, and after pregnancies ending in live births. Am J Psychiatry. 2007 Oct;164(10):1515-20. doi: 10.1176/appi.ajp.2007.06111893. PMID 17898342
- [Background] Marcus SM, Heringhausen JE. Depression in childbearing women: when depression complicates pregnancy. Prim Care. 2009 Mar;36(1):151-65, ix. doi: 10.1016/j.pop.2008.10.011. PMID 19231607
- [Background] Meltzer-Brody S, Boschloo L, Jones I, Sullivan PF, Penninx BW. The EPDS-Lifetime: assessment of lifetime prevalence and risk factors for perinatal depression in a large cohort of depressed women. Arch Womens Ment Health. 2013 Dec;16(6):465-73. doi: 10.1007/s00737-013-0372-9. Epub 2013 Aug 1. PMID 23904137
- [Background] Mian AI. Depression in pregnancy and the postpartum period: balancing adverse effects of untreated illness with treatment risks. J Psychiatr Pract. 2005 Nov;11(6):389-96. doi: 10.1097/00131746-200511000-00005. PMID 16304507
- [Background] Davalos DB, Yadon CA, Tregellas HC. Untreated prenatal maternal depression and the potential risks to offspring: a review. Arch Womens Ment Health. 2012 Feb;15(1):1-14. doi: 10.1007/s00737-011-0251-1. Epub 2012 Jan 4. PMID 22215285
- [Background] Anderson G, Maes M. Postpartum depression: psychoneuroimmunological underpinnings and treatment. Neuropsychiatr Dis Treat. 2013;9:277-87. doi: 10.2147/NDT.S25320. Epub 2013 Feb 21. PMID 23459664
- [Background] Groer MW, Morgan K. Immune, health and endocrine characteristics of depressed postpartum mothers. Psychoneuroendocrinology. 2007 Feb;32(2):133-9. doi: 10.1016/j.psyneuen.2006.11.007. Epub 2007 Jan 3. PMID 17207585
- [Background] Jolley SN, Elmore S, Barnard KE, Carr DB. Dysregulation of the hypothalamic-pituitary-adrenal axis in postpartum depression. Biol Res Nurs. 2007 Jan;8(3):210-22. doi: 10.1177/1099800406294598. PMID 17172320
- [Background] Koleva H, Stuart S, O'Hara MW, Bowman-Reif J. Risk factors for depressive symptoms during pregnancy. Arch Womens Ment Health. 2011 Apr;14(2):99-105. doi: 10.1007/s00737-010-0184-0. Epub 2010 Sep 25. PMID 20872153
- [Background] Meltzer-Brody S. Mental illness is prevalent among U.K. women in the perinatal period and is associated with socioeconomic deprivation. Evid Based Ment Health. 2013 May;16(2):57. doi: 10.1136/eb-2013-101226. Epub 2013 Mar 16. No abstract available. PMID 23503977
- [Background] Arck PC, Hecher K. Fetomaternal immune cross-talk and its consequences for maternal and offspring's health. Nat Med. 2013 May;19(5):548-56. doi: 10.1038/nm.3160. Epub 2013 May 7. PMID 23652115
- [Background] Rowe JH, Ertelt JM, Xin L, Way SS. Regulatory T cells and the immune pathogenesis of prenatal infection. Reproduction. 2013 Oct 21;146(6):R191-203. doi: 10.1530/REP-13-0262. Print 2013 Dec. PMID 23929902
- [Background] Honig A, Rieger L, Kapp M, Sutterlin M, Dietl J, Kammerer U. Indoleamine 2,3-dioxygenase (IDO) expression in invasive extravillous trophoblast supports role of the enzyme for materno-fetal tolerance. J Reprod Immunol. 2004 Apr;61(2):79-86. doi: 10.1016/j.jri.2003.11.002. PMID 15063631
- [Background] Zhu BT. Development of selective immune tolerance towards the allogeneic fetus during pregnancy: Role of tryptophan catabolites (Review). Int J Mol Med. 2010 Jun;25(6):831-5. doi: 10.3892/ijmm_00000411. PMID 20428785
- [Background] Manuelpillai U, Ligam P, Smythe G, Wallace EM, Hirst J, Walker DW. Identification of kynurenine pathway enzyme mRNAs and metabolites in human placenta: up-regulation by inflammatory stimuli and with clinical infection. Am J Obstet Gynecol. 2005 Jan;192(1):280-8. doi: 10.1016/j.ajog.2004.06.090. PMID 15672037
- [Background] Lindqvist D, Janelidze S, Hagell P, Erhardt S, Samuelsson M, Minthon L, Hansson O, Bjorkqvist M, Traskman-Bendz L, Brundin L. Interleukin-6 is elevated in the cerebrospinal fluid of suicide attempters and related to symptom severity. Biol Psychiatry. 2009 Aug 1;66(3):287-92. doi: 10.1016/j.biopsych.2009.01.030. Epub 2009 Mar 6. PMID 19268915
- [Background] Janelidze S, Mattei D, Westrin A, Traskman-Bendz L, Brundin L. Cytokine levels in the blood may distinguish suicide attempters from depressed patients. Brain Behav Immun. 2011 Feb;25(2):335-9. doi: 10.1016/j.bbi.2010.10.010. Epub 2010 Oct 15. PMID 20951793
- [Background] Erhardt S, Lim CK, Linderholm KR, Janelidze S, Lindqvist D, Samuelsson M, Lundberg K, Postolache TT, Traskman-Bendz L, Guillemin GJ, Brundin L. Connecting inflammation with glutamate agonism in suicidality. Neuropsychopharmacology. 2013 Apr;38(5):743-52. doi: 10.1038/npp.2012.248. Epub 2012 Dec 3. PMID 23299933
- [Derived] Sha Q, Madaj Z, Keaton S, Escobar Galvis ML, Smart L, Krzyzanowski S, Fazleabas AT, Leach R, Postolache TT, Achtyes ED, Brundin L. Cytokines and tryptophan metabolites can predict depressive symptoms in pregnancy. Transl Psychiatry. 2022 Jan 26;12(1):35. doi: 10.1038/s41398-022-01801-8. PMID 35078975
- See also: Van Andel Institutes — http://www.vai.org
- See also: Pine Rest Christian Mental Health Services — http://www.pinerest.org